CLINICAL TRIAL: NCT01211990
Title: An Exploratory Study of the Characteristics of and Challenges for International Families Seeking Medical Care in the United States
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100192; 10-M-0192
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-05-13

CONDITIONS: Cancer; Allogeneic Peripheral Blood Stem Cell Transplant; Bone Marrow Transplantation
Keywords: Pediatric; Children; Cancer; Bone Marrow Transplant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- State-of-the art care for children with cancer or rare diseases is not available in all countries. Owing to the proximity of Latin America and the growing numbers of Latinos already in the United States, many international patients receiving specialized medical care in U.S. hospitals are from Spanish-speaking countries. Although there are benefits associated with obtaining specialized care in the United States, linguistic barriers and cultural differences as well as the general stresses of caring for a child with a serious illness may affect families ability to obtain adequate care for their children. Researchers are interested in exploring the experiences and needs of international Latino families receiving medical care for their child in the United States in order to help health care centers provide more appropriate resources and improve the overall quality of culturally sensitive care.

Objectives:

- To understand the experiences of international Latino families who are receiving treatment for their child or have enrolled their child in a research study in the United States.

Eligibility:

* Caregivers of a child between birth and 25 years of ages who are from Latin America (which includes Mexico, all countries in Central America and South America, and Spanish-speaking Caribbean countries) and who have traveled to the United States to enroll their child in a research protocol and/or seek treatment for their child s medical condition.
* Caregivers must have a child enrolled on a research protocol at the time of this study.
* Caregivers must have been away from their country of origin for a minimum of 3 months.

Design:

* This study requires a single interview that should take approximately 1 hour.
* Participants will complete the interview with a member of the research team who is bilingual or fluent in Spanish.
* Participants will be asked open-ended questions about why they chose to come to the United States, how they are adjusting to living and getting medical care for their child in the United States, and what hopes they have for treatment outcomes and future medical care.
* Researchers will record the interviews to be reviewed later. The recordings will be used for this study only.

DETAILED DESCRIPTION:
Background:

The number of individuals who choose to travel out of their native country for medical treatment in the United States has been growing (Purnell & Paulanka, 1998). State-of-the art care for children with cancer or rare diseases is not available in all countries, especially those where the ubiquity of cancer is a new phenomenon (Granda-Cameron, 1999). Due to the proximity of Latin America and the growing numbers of Latinos already in the United States, many, though not all, of the international patients being treated in U.S. hospitals are from Spanish-speaking countries (Coatsworth, Duncan, Pantin, & Szapocznik, 2006). While there are benefits associated with obtaining care in the United States such as improved access to specialized medical services, barriers posed by linguistic and cultural differences may play a role in the provision of adequate care for these children and their families. Additional challenges associated with receiving care in another country include failure to adhere to medical regimen due to breakdowns in communication, increased stress upon the caregiver to navigate a foreign health system and adjust to a foreign culture, and being uprooted from supportive social networks and family members (Flores, Abreu, Schwartz, & Hill, 2000). Parents of children with more severe and/or complex diseases may find themselves settling in the United States at the cost of leaving behind loved ones and careers in their country of origin. Provision of optimal care for these patients includes addressing the adjustment needs of their families; the caregiver-patient relationship has a significant influence on the child s physical and psychological outcomes (Brown et al., 2008). Exploring the experiences and needs of internationalfamilies that come to the United States seeking medical care for their child may help health care centers to provide more appropriate resources and may improve the overall quality of culturally-sensitive care provided to these families.

Objective: This is a pilot, exploratory study designed to obtain greater understanding about the unique experiences of international families, mostly Latino families, who choose to participate in clinical research or seek medical treatment in the United States. Due to the lack of research on this phenomenon, the study will utilize qualitative methods to extrapolate the main themes that characterize this experience. The end goal of the study is to identify unique risk and protective factors that link directly to feasible interventions, so that we can provide this growing population with the standard of care expected by the mission of the NIH.

Aims:

To identify factors affecting the decision by international caregivers to seek treatment in the United States, with a specific focus on how medical information is obtained and utilized in the decision-making process.

To explore the experience of international caregivers in adapting to the medical and social culture of the United States.

To explore the thoughts and concerns of international caregivers regarding termination of treatment and subsequent re-entry into their native country.

To identify the presence and kind of positive growth experiences that occur in international families seeking medical care in the United States

To develop a set of concrete risk and protective factors associated with this experience in order to link to feasible interventions.

(The term caregiver in this protocol is used to encapsulate any individual, such as a parent, close relative, foster parent, or head of household, who attends to the needs of the ill child.)

Study Population:

This is a study taking place at the National Institutes of Health (NIH). All caregivers of a child between the ages of 0-25 from a foreign country who have traveled to the United States for the purpose of enrolling in a research protocol and/or seeking treatment for their child s medical condition will be invited to participate in this study. Caregivers who immigrated to the United States for reasons other than obtaining these services for their child s condition will not be eligible to enroll in this study. Given the present demographic populations at NIH, it is expected that participants will include, but not be limited to, individuals from the Caribbean, Dominican Republic, Puerto Rico, Chile, Peru, Guatemala, and Mexico. This sampling frame ensures that the presence of black, white, and mixed race individuals will be represented, acknowledging ethnicities that are often overlooked in studies focusing specifically on the experience of a given ethnic or racial group.

Socioeconomic situation of the families is expected to vary widely; at NIH, individuals who meet the criteria for this study are from all different socioeconomic strata and have varying levels of education.

Design:

This is a qualitative study that will utilize narrative interview techniques to gather data, and content analysis techniques to analyze data. Data will be gathered according to theories of saturation of content, while collecting sufficient data to ensure credibility and face validity (Mays & Pope, 2000). NVivo, a validated quantitative research tool will be used for data analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Caregivers of children aged 0-25.
* The children of the participants must be involved in clinical research or be receiving treatment for their child s medical condition. This includes but is not limited to oncological and hematological diseases, conditions requiring transplant, and rare immunodeficiency or genetic conditions.
* The family traveled to the US for the purpose of addressing their child s medical condition.
* Caregivers must be from a country outside of the United States. Care givers must be fluent in Spanish or English.
* Caregiver has been away from the country of origin for a minimum of three months.
* The child s treatment protocol PI must agree to have the research team contact potential participants in order to explore their interest in this protocol.

EXCLUSION CRITERIA:

* The caregiver participant immigrated to the US for reasons other than enrolling in a research study or addressing their child s medical condition.
* Presence of psychotic symptoms or severe psychological distress, which in the judgment of the Principal or Associate Investigator or consulting psychiatrist would compromise the caregiver s ability to engage in the interview or is likely to interfere with the study procedures or results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-08-31; Study Completion 2013-05-13

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbe M, Simon C, Angiolillo A, Ruccione K, Kodish ED. A survey of language barriers from the perspective of pediatric oncologists, interpreters, and parents. Pediatr Blood Cancer. 2006 Nov;47(6):819-24. doi: 10.1002/pbc.20841. PMID 16615062
- [Background] Alegria M, Canino G, Rios R, Vera M, Calderon J, Rusch D, Ortega AN. Inequalities in use of specialty mental health services among Latinos, African Americans, and non-Latino whites. Psychiatr Serv. 2002 Dec;53(12):1547-55. doi: 10.1176/appi.ps.53.12.1547. PMID 12461214
- [Background] Barakat LP, Kazak AE, Meadows AT, Casey R, Meeske K, Stuber ML. Families surviving childhood cancer: a comparison of posttraumatic stress symptoms with families of healthy children. J Pediatr Psychol. 1997 Dec;22(6):843-59. doi: 10.1093/jpepsy/22.6.843. PMID 9494321